CLINICAL TRIAL: NCT06910540
Title: Acupuncture-type Transcutaneous Electrical Nerve Stimulation on Pain and Stress Reduction Before and During Transvaginal Ultrasound-guided Oocyte Retrieval: a Randomized Controlled Trial
Brief Title: ACU-TENS on Pain and Stress Reduction Before and During TUGOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025.106
Record Dates: First submitted 2025-03-26; First posted 2025-04-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Oocyte Retrieival and Post Operative Pain Control; Acupuncture
Keywords: Transvaginal ultrasound-guided oocyte retrieval; Acupuncture-type transcutaneous electrical nerve stimulation; Pain control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acu-TENS (Experimental): Acu-TENS treatment
  Interventions: Other: Acu-TENS
- Sham acu-TENS (Sham Comparator): Sham acu-TENS without electric current
  Interventions: Other: Sham acu-TENS

INTERVENTIONS:
Other: Acu-TENS — This protocol makes use of the acu-TENS treatment on the acupoints Hegu (LI4), Zusanli (ST36), Sanyinjiao (SP6), and Taichong (LR3). After cleaning the acupoints with alcohol, electrode pads (HC-ROUND-32 2.0) will be placed on the acupoints according to the locations described in the Standard International Acupuncture Nomenclature. The electrode pads will be connected to a TENS machine (MTR+ Myolito Multifunctional Stimulator MTRP-00003), in which ipsilateral LI4 and SP36, SP6 and LR3 serve a pair. A pulse rate of 120 Hz, current of 3-5 mA, and pulse width of 300µS will be delivered continually during TUGOR.
  Arms: Acu-TENS
Other: Sham acu-TENS — In the sham acu-TENS, within the same time interval, TENS pads will be placed on the same acupoints, connected to the machine, but without electric current.
  Arms: Sham acu-TENS

SUMMARY:
Objectives: To demonstrate the use of acupuncture-type transcutaneous electrical nerve stimulation (acu-TENS) during transvaginal ultrasound-guided oocyte retrieval (TUGOR) will reduce 50% of the intensity of pain experienced by women.

Hypothesis to be tested: Does the use of acu-TENS reduce 50% of pain in TUGOR? Design and subjects: A prospective randomized control trial will be carried out at the Department of Obstetrics and Gynaecology, Prince of Wales Hospital. 144 women undergoing TUGOR will be randomized to receive acu-TENS or sham acu-TENS for pain control during TUGOR.

Study instruments: During the TUGOR procedure, ultrasound of the pelvis will be performed by Aloka ProSound SSD-3500SX device (Japan). Each follicle will be pierced using a single lumen ovum aspiration needle or a double lumen ovum aspiration catheter (COOK Medical, UK) under ultrasound guidance. Acu-TENS will be done using MTR+ Myolito Multifunctional Stimulator.

Main outcome measures: Primary outcome is the pain score before and during TUGOR. Secondary outcomes include (1) other pain level parameters including pain control satisfaction, surgeon's assessment of the patient co-operation score and patient intraoperative pain; (2) stress and anxiety levels, Stait Trait Anxiety Inventory, General Health Questionnaire, Beck Depression Inventory, and saliva cortisol; (3) patient's satisfaction measured by Client Satisfaction Questionnaire and satisfaction score on pain control; (4) difficulty in retrieving oocytes; (5) IVF parameters; (6) safety profile; and (7) bias assessment.

Data analysis: Data analysis will be performed using Statistical Packages of Social Sciences for Windows.

Expected results: The investigators expect that acu-TENS will reduce 50% of pain in TUGOR.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF-ET cycles are to be recruited from the Assisted Reproduction Technology unit in the Prince of Wales Hospital

Exclusion Criteria:

* Patient not eligible for acu-TENS
* Patient with severe cardiac and respiratory disease history
* Smoker or drinker
* Refuse or incompetence for informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain VAS (minimum 0 to maximum 100) | Before admission and 1 hour before TUGOR, when switch to contra-lateral ovary, shortly after TUGOR, and 30 minutes, 1 hour, 2 hours, and 4 hours after TUGOR
  Research assistance who is not involved in the TUGOR will ask patients about the pain level by a ruler on 100mm visual analogous scale (VAS; 0 mm = no pain, 100mm = worst pain). Before operation, patient will be asked to give VAS pain and anxiety before admission and 1 hour before TUGOR. This is to assess the baseline pain perception for the patients. VAS for vaginal and abdominal pain and will be rated by patient when the surgeon switch to contra-lateral ovary and shortly after TUGOR. Patient will be asked to rate the abdominal and vaginal pain again 30 minutes, 1 hour, 2 hours, and 4 hours after TUGOR (before discharge). With a change of more than or equal to 10 for the 100 mm VAS, the analgesic intervention is clinical important.

SECONDARY OUTCOMES:
Satisfaction score (minimum 0 to maximum 100) | 4 hour after TUGOR
  Patient will be asked to give the satisfaction score regarding the pain control of TUGOR: excellent, satisfactory, fair and unsatisfactory. For those patients had undergone previous oocyte retrieval by conscious sedation alone, they will ask whether they prefer the present treatment modality or not.
Patient compliance index (minimum 1 to maximum 5) | 4 hour after TUGOR
  To validate the VAS pain score rated by patients, surgeons will rate the patient compliance index. For the patient compliance index, it is a 5-point Likert scale rated from 1 (fully co-operation) to 5 (no co-operation, procedure abandoned).
Patient pain score (minimum 0 to maximum 4) | 4 hour after TUGOR
  To validate the VAS pain score rated by patients, surgeons will rate the patient pain score. For the patient pain score, it is a 5-point Likert scale rated from 0 (patient did not show any sign of pain) to 4 (patient did not let the procedure continue which was demonstrated by verbal or bodily expression).
Additional use of analgesia | 4 hour after TUGOR
  The additional of analgesic during and after TUGOR will be recorded.
Spielberger's State Anxiety Inventory (minimum 20 to maximum 80) | Before admission and 1 hour after TUGOR
  Basal anxiety level will be assessed by the Spielberger's State Anxiety Inventory (STAI; both the S-AD questionnaire for stress level and T-AI questionnaire for traits). As stress state may affect the pain level, S-AD questionnaire will be done again after TUGOR.
12-item General Health Questionnaire (minimum 12 to maximum 48) | Before admission.
  Basal anxiety level will be assessed by the 12-item General Health Questionnaire (GHQ-12).
Beck Depression Inventory (minimum 0 to maximum 63) | Before admission.
  Basal anxiety level will be assessed by the Beck Depression Inventory (BDI).
Saliva cortisol | Before admission and 1 hour after TUGOR
  Saliva cortisol would be utilized as an objective indicator of our patient's stress level while undergoing TUGOR. Saliva cortisol will be measured before and immediately after TUGOR procedures.
Number of participants with treatment-related adverse events | Before admission.
  Patients will be invited to try on the TENS pads to see if they are allergic to it. This will be assessed by observing if their skin may become red and irritated.
  Any treatment-related dizziness, headache, tiredness will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Pui Wah, Jacqueline, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided